CLINICAL TRIAL: NCT00113373
Title: A Phase II Evaluation of Lapatinib (GW572016) (NCI-Supplied Agent, NSC #727989) in the Treatment of Persistent or Recurrent Epithelial Ovarian or Primary Peritoneal Carcinoma
Brief Title: Lapatinib in Treating Patients With Persistent or Recurrent Ovarian Epithelial or Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02654; NCI-2012-02654 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000429548; GOG-0170G (Other: Gynecologic Oncology Group); GOG-0170G (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine

ARMS (1):
- Treatment (lapatinib ditosylate) (Experimental): Patients receive oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lapatinib ditosylate — Given orally
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. This phase II trial is studying how well lapatinib works in treating patients with persistent or recurrent ovarian epithelial or peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: Primary I. Determine 6-month progression-free survival of patients with persistent or recurrent ovarian epithelial or primary peritoneal cancer treated with lapatinib.

II. Determine the nature and degree of toxicity of this drug in these patients.

Secondary I. Determine the clinical response rate (partial and complete response) in patients treated with this drug.

II. Determine the duration of progression-free and overall survival of patients treated with this drug.

III. Determine the impact of prognostic variables, including platinum sensitivity, performance status, and cellular histology (clear cell or mucinous type), on patients treated with this drug.

IV. Correlate tumor levels of expression of epidermal growth factor receptors (EGFR), phosphorylated EGFR, HER2/neu, and Ki-67, as determined by immunohistochemistry, with clinical response in patients treated with this drug.

V. Correlate EGFR mutations in tumor DNA with clinical response in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 22-60 patients will be accrued for this study within 12-26 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed persistent or recurrent ovarian epithelial or primary peritoneal cancer
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
  * Presence of ≥ 1 target lesion

    * Tumors within a previously irradiated field are not considered target lesions unless evidence of progression is documented or proven by biopsy 3 months after completion of radiotherapy
* Disease progression during OR persistent disease after 1 prior platinum-based chemotherapy regimen* for primary disease containing carboplatin, cisplatin, or another organoplatinum compound

  * Initial treatment may have included high-dose therapy, consolidation therapy, or extended therapy administered after surgical or non-surgical assessment
  * Treatment-free interval after platinum-based chemotherapy < 12 months
* Tumor accessible by guided core needle or fine needle biopsy
* Ineligible for any higher priority Gynecologic Oncology Group (GOG) protocols (i.e., any active phase III protocol for the same patient population)
* Performance status - GOG 0-2 (patients who have received 1 prior treatment regimen)
* Performance status - GOG 0-1 (patients who have received 2 prior treatment regimens)
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Serum Glutamate Oxaloacetate Transaminase (SGOT) ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Ejection fraction normal by echocardiogram or MUGA
* No GI disease resulting in an inability to take oral medication
* No malabsorption syndrome
* No requirement for IV alimentation
* No uncontrolled inflammatory GI disease (e.g., Crohn's disease or ulcerative colitis)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 1 month after completion of study treatment
* No active infection requiring antibiotics
* No sensory or motor neuropathy > grade 1
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to lapatinib
* At least 4 weeks since prior immunologic agents for the malignancy
* No prior trastuzumab (Herceptin®)or cetuximab
* See Disease Characteristics
* Recovered from prior chemotherapy
* At least 6 weeks since prior nitrosoureas or mitomycin for the malignancy
* No prior non-cytotoxic chemotherapy for recurrent or persistent disease
* At least 2 weeks since prior and no concurrent dexamethasone or dexamethasone equivalent dose > 1.5 mg/day
* At least 1 week since prior hormonal therapy for the malignancy
* Concurrent hormone replacement therapy allowed
* See Disease Characteristics
* Recovered from prior radiotherapy
* No prior radiotherapy to > 25% of marrow-bearing areas
* See Disease Characteristics
* Recovered from prior surgery
* No prior surgical procedure affecting gastrointestinal (GI) absorption
* At least 4 weeks since other prior therapy for the malignancy
* At least 6 months since prior and no concurrent amiodarone
* At least 1 week since other prior and no concurrent CYP3A4 inhibitors
* At least 2 weeks since prior and no concurrent CYP3A4 inducers
* At least 1 week since prior and no concurrent H2 inhibitors or proton pump inhibitors

  * Concurrent antacids allowed provided they are not administered within 1 hour before and 1 hour after study drug administration
* No prior cancer treatment that would preclude study treatment
* No prior lapatinib
* No other prior target-specific therapy directed to the HER family (e.g., gefitinib or erlotinib)
* No concurrent herbal medications
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 5/2/2005 and closed to accrual on 5/1/2006.
Groups:
- Lapatinib: 1500 mg of lapatinib orally every day (cycle = 28 days) until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | Lapatinib
Started | 28
Completed | 25 (Eligible and treated patients.)
Not Completed | 3
Not completed — Ineligible: wrong primary | 1
Not completed — Ineligible: second primary | 1
Not completed — Never Treated | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients.
Arm/Group | Lapatinib
Number analyzed (Participants) | 25
Age, Continuous [Median (Standard Deviation); unit: years] | 63.4 (9.3)
Age, Customized [Number; unit: participants]
  40-49 years | 3
  50-59 years | 4
  60-69 years | 12
  70-79 years | 4
  80-89 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
International Federation of Gynecology and Obstetrics (FIGO) Stage Recurrent/Persistent [Number; unit: participants] | 25
Histologic Type [Number; unit: participants]
  Endometrioid Adenocarcinoma | 3
  Undifferentiated Carcinoma | 2
  Serous Adenocarcinoma | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) > 6 Months
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: For those patients whose disease can be evaluated by physical examination, progression was assessed prior to each 28-day cycle. CT scan or MRI if used to follow measurable disease every other cycle for the first 6 months
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lapatinib
Number analyzed (Participants) | 25
percentage of participants | 8.0 [1.4 to 23.1]

2. Primary Outcome: Frequency and Severity of Adverse Effects as Assessed by Common Toxicity Criteria for Adverse Events (CTCAE) v3.0
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment
Population: Eligible and evaluable
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 3.0
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 3.0
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 3.0
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 3.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0)
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
Participants
  Leukopenia | 23 | 2 | 0 | 0 | 0
  Thrombocytopenia | 24 | 1 | 0 | 0 | 0
  Anemia | 12 | 10 | 3 | 0 | 0
  Other hematologic | 24 | 1 | 0 | 0 | 0
  Hearing | 21 | 0 | 4 | 0 | 0
  Constitutional | 12 | 9 | 1 | 2 | 1
  Dermatologic | 15 | 6 | 4 | 0 | 0
  Gastrointestinal | 5 | 11 | 5 | 4 | 0
  Hemorrhage | 23 | 2 | 0 | 0 | 0
  Infection | 24 | 0 | 1 | 0 | 0
  Lymphatics | 24 | 1 | 0 | 0 | 0
  Musculoskeletal | 22 | 1 | 1 | 1 | 0
  Metabolic | 13 | 8 | 2 | 2 | 0
  Neuropathy | 21 | 2 | 1 | 1 | 0
  Ocular | 24 | 1 | 0 | 0 | 0
  Pain | 17 | 7 | 0 | 1 | 0
  Pulmonary | 23 | 2 | 0 | 0 | 0

3. Secondary Outcome: Tumor Response
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: Baseline, every other cycle for 6 months and then every 6 months for up to 5 years
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lapatinib
Number analyzed (Participants) | 25
percentage of participants | 0 [0.0 to 8.8]

4. Secondary Outcome: Duration of Progression-free Survival
Description: as for outcome 1
Time Frame: Every other cycle for 6 months and then every 6 months for up to 5 years.
Population: Eligible and evaluable patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib
Number analyzed (Participants) | 25
months | 1.77 [1.28 to 1.87]

5. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or the date of last contact.
Time Frame: From entry into the study to death or the date of last contact, assessed up to 5 years
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib
Number analyzed (Participants) | 25
months | 10.5 [3.4 to 17.0]

6. Secondary Outcome: Prognostic Variable: Platinum Sensitivity
Description: Patients who had disease progression within 6 months of ending their last regimen of platinum therapy were considered platinum resistant. Patients who had disease progression between 6 and 12 months of ending their last platinum regimen were considered platinum sensitive. Patients who had disease progression beyond12 months of ending their last platinum regimen were also considered platinum sensitive.
Time Frame: Baseline
Population: Eligible and evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib
Number analyzed (Participants) | 25
Participants
  Platinum Sensitive | 9
  Platinum Resistant | 16

7. Secondary Outcome: Prognostic Variables: Performance Status
Description: Performance Status 0 = Fully active, able to carry on all pre-disease performance without restriction Performance Status 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature, e.g., light housework, office work Performance Status 2 = Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours.
Time Frame: Baseline
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib
Number analyzed (Participants) | 25
Participants
  Performance Status 0 | 18
  Performance Status 1 | 6
  Performance Status 2 | 1

8. Secondary Outcome: Prognostic Variable: Cellular Histology
Description: Number of patients with Clear Cell Carcinoma or Mucinous Carcinoma
Time Frame: Baseline
Population: Eligible and evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib
Number analyzed (Participants) | 25
Participants
  Clear Cell Carcinoma | 0
  Mucinous Carcinoma | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are all Serious Adverse Events (SAEs) for up to 5 years after stopping study treatment
Arm/Group | Lapatinib
Serious Adverse Events (participants affected / at risk) | 10/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib (N=25)
Death No Ctcae Term - Disease Progression Nos (General disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 1
Death No Ctcae Term - Death Nos (General disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib (N=25)
Tinnitus (Ear and labyrinth disorders) | 4
Platelets (Blood and lymphatic system disorders) | 1
Leukocytes (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 15
Hypertension (Cardiac disorders) | 2
Sweating (General disorders) | 1
Weight Loss (General disorders) | 2
Fatigue (General disorders) | 13
Death No Ctcae Term - Death Nos (General disorders) | 1
Nail Changes (Skin and subcutaneous tissue disorders) | 1
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 4
Acne (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2
Hand-Foot (Skin and subcutaneous tissue disorders) | 1
Hot Flashes (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Distention (Gastrointestinal disorders) | 4
Taste Alteration (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 7
Anorexia (Gastrointestinal disorders) | 5
Dehydration (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 16
Diarrhea (Gastrointestinal disorders) | 18
Hemorrhage, Gu - Vagina (Vascular disorders) | 2
Hemorrhage, Gi - Rectum (Vascular disorders) | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 3
Hemorrhage, Gu - Bladder (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 1
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 1
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 1
Edema: Limb (Blood and lymphatic system disorders) | 2
Ast (Metabolism and nutrition disorders) | 3
Cholesterol,serum High (Metabolism and nutrition disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Alt (Metabolism and nutrition disorders) | 3
Alkaline Phosphatase (Metabolism and nutrition disorders) | 3
Bilirubin (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 6
Hyperuricemia (Metabolism and nutrition disorders) | 1
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Soft Tissue Necrosis - Abdomen (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Joint-Function (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 1
Mood Alteration - Depression (Nervous system disorders) | 7
Mood Alteration - Anxiety (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Neuropathy-Sensory (Nervous system disorders) | 5
Flashing Lights/Floaters (Eye disorders) | 1
Pain: Pelvis (General disorders) | 1
Pain: Vagina (General disorders) | 1
Pain: Head/Headache (General disorders) | 4
Pain: Extremity-Limb (General disorders) | 1
Pain: Back (General disorders) | 1
Pain: Joint (General disorders) | 1
Pain: Bladder (General disorders) | 1
Pain: Stomach (General disorders) | 2
Pain: Oral Cavity (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 10
Pain: Muscle (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Bladder Spasm (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 2

LIMITATIONS AND CAVEATS:
The clinical trial was a two-stage design, accruing approximately 25 patients in each stage. Early termination of the study would result if warranted from an interim futility analysis. This study stopped early for lack of treatment efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less